CLINICAL TRIAL: NCT00955565
Title: Accuracy of Navigation in Placement of Sacroiliac Screw. Multicenter Randomized Controlled Trial
Brief Title: Accuracy of Navigation in Placement of Sacroiliac Screw
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Ulrich C. Stöckle, Klinikum rechts der Isar der TU München
Organization: AO Innovation Translation Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sacroliac screw-08
Record Dates: First submitted 2009-07-17; First posted 2009-08-10 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Navigated (Experimental)
  Interventions: Procedure: Navigated
- Conventional (Active Comparator)
  Interventions: Procedure: Conventional

INTERVENTIONS:
Procedure: Navigated — Subjects receive receive computer assisted placement of the sacroiliac screws. The computer assisted placement will be performed by using the BrainLab Vector Vision®Trauma Navigation Software. Two approaches will be used, the 2D navigation and 3D navigation.
  Other Names: BrainLab Vector Vision®Trauma Navigation Software
  Arms: Navigated
Procedure: Conventional — Subjects receive standard fluoroscopic placement of the sacroiliac screw.
  Arms: Conventional

SUMMARY:
The purpose of this study is to compare the precision of computer-assisted navigation for hip screw implantation to conventional fixation without navigation.

DETAILED DESCRIPTION:
Standard treatment for sacroiliac dislocations and sacroiliac fractures is placement of two screws through the iliosacral joint into the sacral ala or the body of the S1 vertebra. Correct positioning is technically demanding. Screw displacement may reduce the strength of fixation and lead to neurological complications.

Secondary objectives of the study are to compare the fluoroscopy time, complications and surgery duration between the treatments.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically confirmed sacroiliac dislocation or sacroiliac fracture
* Sacroiliac arthritis
* Age 18 years and more
* Written informed consent by patient or his/her legal representative

Exclusion Criteria:

* Poor life expectancy (<3months)
* Fracture of pathologic origin
* History of substance abuse (recreational drugs, alcohol)within 12 months prior to screening
* Prisoner
* Currently involved in another study that precludes or complicates participation
* Disease or condition that would preclude accurate evaluation (e.g., significant psychiatric disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Proportion of misplaced sacroiliac screws as evaluated by postop CT-scanning. | 2 days

SECONDARY OUTCOMES:
Fluoroscopic time, complications and surgery duration. | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Beate P. Hanson, MD, Study Director — AO Clinical Investigation and Documentation, Davos, Switzerland; Ulrich C. Stöckle, Prof. MD, Principal Investigator — Klinikum rechts der Isar der TU München
Locations (9):
- University of Virginia Health System, Charlottesville, Virginia, United States
- Germany (7):
  - Charité Berlin, Campus Virchow Klinikum, Berlin
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum des Saarlandes, Homburg
  - Klinikum rechts der Isar der TU München, München
  - Universitätsklinikum Münster, Münster
  - Katharinenhospital, Stuttgart
  - Universität Ulm, Ulm
- Rashid Hospital, Dubai, United Arab Emirates